CLINICAL TRIAL: NCT06770075
Title: Brightline - a Digital Phenotyping Study Toward Advancing Mental Health on Campus
Brief Title: Brightline: Advancing Mental Health on Campus
Status: Recruiting | Type: Observational
Sponsor: Nanyang Technological University (Other)
Collaborators: MOH Office for Healthcare Transformation (MOHT), Singapore (Unknown)
Responsible Party: Principal Investigator, Andy Khong W H, Assoc Prof, Nanyang Technological University
Other Study IDs: IRB-2023-894
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Depression; Anxiety; Stress; Positive Affect; Negative Affect; Loneliness
Keywords: university student; mental health; digital phenotyping; digital biomarkers; passive sensing; risk prediction; mental health seeking
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Undergraduate students: Undergraduate students from Nanyang Technological University
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Participants will not receive any study intervention. During the six month study period, participants will complete four active assessments at Months 0, 1, 3 and 6, and data from the study-provided wearable (Fitbit Charge 6) and sensors from the participant's smartphone (through the Brightline app) will be collected passively throughout.
  Other Names: There will be no interventions involved in this study.

SUMMARY:
This observational study will employ a multi-modal observation methodology, integrating data from wearable devices and smartphones to establish comprehensive digital biomarkers for identifying symptoms of mental health conditions in university students. The study aims to identify the digital behavioural markers associated with mental health conditions, develop predictive algorithms for mental health states from digital markers, and identify university students at risk for mental health conditions.

DETAILED DESCRIPTION:
In this study, participants will be monitored over a six-month period to determine the association between digital behavioural markers and mental health symptoms among university students. Participants will be passively monitored to collect digital phenotyping data (e.g., physical activity, sleep activity, heart rate, physiological patterns, sociability indices, finger taps, ambient light, phone states, etc.), using a wearable device and sensors from the smartphone. Participants will also complete self-report questionnaires at Months 0, 1, 3, and 6, to track changes in mental health symptoms and behavioural data. The collected data will be analysed to examine the longitudinal changes in depression, anxiety, and other mental health issues among university students and explore the feasibility of data collection procedures.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 years or older.
* Be a current full-time undergraduate student.
* Own a smartphone with Wi-Fi, 4G, and Bluetooth capabilities.
* Possess adequate English language proficiency.
* Be able to download the study apps.
* Provide informed consent.

Exclusion Criteria:

* Are part-time students.
* Have a current diagnosis of any mental health disorder or a past diagnosis with any bipolar disorder, substance use disorder, or any psychotic disorder.
* Are currently undergoing mental health treatment.
* Lack sufficient English proficiency.
* Report suicidal ideation as indicated by Patient Health Questionnaire (PHQ-9) Item-9, "Thoughts you would be better off dead or of hurting yourself in some way".
* Cannot commit to wearing a wearable device for the six-month monitoring period.
* Receive special education accommodations or support from the university.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Undergraduate students
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline (Month 0), Interim (Month 1), Mid-point (Month 3), End-point (Month 6)
  A nine-item scale assessing depression severity. A higher total score indicates increased depression severity.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Baseline (Month 0), Interim (Month 1), Mid-point (Month 3), End-point (Month 6)
  A seven-item scale assessing anxiety severity. A higher total score indicates increased anxiety severity.
Perceived Stress Scale 4 (PSS-4) | Baseline (Month 0), Interim (Month 1), Mid-point (Month 3), End-point (Month 6)
  A four-item scale assessing stress severity. A higher total score indicates increased stress severity.
International Positive and Negative Affect Schedule - Short Form (I-PANAS-SF) | Baseline (Month 0), Interim (Month 1), Mid-point (Month 3), End-point (Month 6)
  A ten-item scale divided into two subscales, assessing subjective experiences of positive and negative affect. A higher total score on each subscale indicates increased positive or negative affect.
University of California Los Angeles, 3-Item Loneliness Scale (UCLA-3) | Baseline (Month 0), Interim (Month 1), Mid-point (Month 3), End-point (Month 6)
  A three-item scale assessing levels of loneliness. A higher total score indicates increased loneliness.
University Stress Scale (USS) | Baseline (Month 0), Interim (Month 1), Mid-point (Month 3), End-point (Month 6)
  A 21-item scale assessing the degree to which university life events are perceived as stressful. A higher score indicates increased perceived stress.
Mental Help Seeking Attitudes Scale (MHSAS) | Baseline (Month 0), End-point (Month 6)
  A nine-item scale assessing attitudes towards seeking mental health help. A higher score indicates more favorable attitudes towards seeking mental health assistance.
Perceptions of study compliance | End-point (Month 6)
  Participants will be evaluated on five items assessing the acceptability of the study procedure, specifically related to wearing the wearable device. Additionally, they will be provided a free-text response to details any difficulties or challenges encountered during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Andy WH Khong, PhD, Principal Investigator — Nanyang Technological University; Andy HY Ho, PhD, EdD, Principal Investigator — Nanyang Technological University
Locations (1):
- Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ito S, Ang CS, Kampman OP, Rokde K, Buddhika T, Heaukulani C, Tan ZW, Dewanti FA, Au EWM, Huan VS, Morris RJ, Khong AWH, Ho AHY. Harnessing digital phenotyping to advance university student mental health (Brightline) in Singapore: study protocol for a prospective observational study. BMJ Open. 2025 Sep 22;15(9):e103652. doi: 10.1136/bmjopen-2025-103652. PMID 40983586